CLINICAL TRIAL: NCT03117153
Title: Effect of a Liquid Toothpaste on Periodontal Disease : a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of a Liquid Toothpaste on Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-A Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DA-5502_301
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Periodontitis; Gingivitis
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA-5502 liquid toothpaste (Experimental): SMFP 760mg, CPC 50mg, tocopherol acetate 10mg, panthenol 100mg, Dipotassium glycyrrhizinate 20mg.
  everyday 3 times for 6 weeks
  Interventions: Other: DA-5502 liquid toothpaste
- placebo (Placebo Comparator): no active ingredients
  everyday 3 times for 6 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Other: DA-5502 liquid toothpaste — 6 weeks study, brush three times daily, liquid toothpaste
  Other Names: DA-5502, Gumguard
  Arms: DA-5502 liquid toothpaste
Other: placebo — same flavor solution, brush three times daily
  Arms: placebo

SUMMARY:
The aim of the present clinical study is to evaluate the efficacy and safety of the novel toothpaste in patients diagnosed with gingivitis and/or periodontitis.

DETAILED DESCRIPTION:
The trial was a randomized, double-blind, placebo-controlled, parallel group, single-center(Department of periodontology, Yonsei University Dental Hospital) study.

98 patients were assessed for eligibility. Since two patients did not meet the inclusion criteria, 96 subjects were randomly assigned to either the test group.The test group was provided a liquid toothpaste and a control group received placebo. At the end of the study, results were analyzed for 87 patients : 42 in the test group and 45 in the control group .

The study protocol requested 4 visits- once every two weeks-of each subjects in the center. At the baseline, subjects were randomly allocated to the test group or the control group. Scaling and tooth brushing instruction were performed and all of the clinical parameters were evaluated. At the 2- and 4-week examinations, clinical parameters of GI, PI were evaluated and at the 6-week examination, all of the clinical parameters were evaluated.

Also, Microbiological quantitative analysis of this procedure was performed at the baseline and 6-week examinations.

ELIGIBILITY:
Inclusion Criteria:

* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
* Initial gingivitis index of 1.1~2.0 as determined by the use of the Loe and Silness Gingival Index.
* Signed Informed Consent Form.

Exclusion Criteria:

* initial plaque index <1.5, gingival index <1.0
* smoker
* Chronic disease (uncontrolled diabetes, liver disease, heart disease, kidney disease..)
* subject who had hemorrhagic medical history or who take antiplatelet agent or anticoagulant
* subject who need antibiotics for preventive administration
* subjects who had preventive treatment or treatment for periodontitis in the last three months
* Use of orthodontic appliances.
* Pregnant women or women who are breast feeding.
* Previous participation in any other clinical trial in the last 30 days
* Judged unsuitable by investigators for other reasons.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2015-02-11 (Actual)

PRIMARY OUTCOMES:
gingival index | 6 week

SECONDARY OUTCOMES:
Plaque index | 6 week
Clinical attachment level | 6 week
Bleeding of probing | 6 week
change of microbial growth | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Sung Kim, Ph.D, Study Director — Department of Periodontology, Research Institute for Periodontal Regeneration, College of Dentistry, Yonsei University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawlinson A, Pollington S, Walsh TF, Lamb DJ, Marlow I, Haywood J, Wright P. Efficacy of two alcohol-free cetylpyridinium chloride mouthwashes - a randomized double-blind crossover study. J Clin Periodontol. 2008 Mar;35(3):230-5. doi: 10.1111/j.1600-051X.2007.01187.x. Epub 2008 Jan 5. PMID 18190554
- [Background] Hu D, Li X, Sreenivasan PK, DeVizio W. A randomized, double-blind clinical study to assess the antimicrobial effects of a cetylpyridinium chloride mouth rinse on dental plaque bacteria. Clin Ther. 2009 Nov;31(11):2540-8. doi: 10.1016/j.clinthera.2009.11.004. PMID 20109998
- [Background] Silva MF, dos Santos NB, Stewart B, DeVizio W, Proskin HM. A clinical investigation of the efficacy of a commercial mouthrinse containing 0.05% cetylpyridinium chloride to control established dental plaque and gingivitis. J Clin Dent. 2009;20(2):55-61. PMID 19591338
- [Background] Charles CA, McGuire JA, Sharma NC, Qaqish J. Comparative efficacy of two daily use mouthrinses: randomized clinical trial using an experimental gingivitis model. Braz Oral Res. 2011 Jul-Aug;25(4):338-44. doi: 10.1590/s1806-83242011000400010. PMID 21860922
- [Background] Hernandez-Cott PL, Elias Boneta A, Stewart B, DeVizio W, Proskin HM. Clinical investigation of the efficacy of a commercial mouthrinse containing 0.05% cetylpyridinium chloride in reducing dental plaque. J Clin Dent. 2009;20(2):39-44. PMID 19591335